CLINICAL TRIAL: NCT00609297
Title: Opioid Titration in the Hospice Setting: Barriers Assessment and Modification of the Model Order Sheet and Protocol Stage 2, Part A
Brief Title: Pain Control in Hospice Patients With Cancer-Related Pain
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0731; VU-VICC-SUPP-0731; VU-VICC-070605
Record Dates: First submitted 2008-02-06; First posted 2008-02-07 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Pain; Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Supportive Care: Alive Hospice Patients with Pain
  Interventions: Other: medical chart review; Other: questionnaire administration; Other: survey administration

INTERVENTIONS:
Other: medical chart review — The Research Nurse will conduct a chart review after the patient's death.
  Other Names: None specified
Other: questionnaire administration — The questionnaires will be completed at the end of week 1, week 2 and week 4.
  Other Names: None Specified
Other: survey administration — Given to patient and caregivers throughout the study
  Other Names: none specified

SUMMARY:
RATIONALE: Gathering information over time about cancer-related pain from patients in a hospice and their caregivers may help doctors learn more about pain control.

PURPOSE: This clinical trial is studying how well standard pain control works in hospice patients with cancer-related pain.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain prospective data describing standard pain management methods and outcomes in the hospice setting.

OUTLINE: Data regarding pain and pain management is obtained from three sources: the patient, the caregiver(s), and the medical records.

* Patient assessment*: At baseline, patients provide demographic data and complete the Pain Assessment Form verbally via interview. The form addresses average pain, worst pain, pain relief, hours in pain, pain-related distress, and barriers to pain control. Patients are asked to rate pain control. Patients also complete the Pain Communication Survey to assess how they communicate with health care providers about their pain. After the baseline assessment is completed, pain is assessed by the research nurse through home visits* 3 times weekly and telephone interviews twice weekly. During each visit or telephone contact, patients are interviewed to complete the Pain Assessment Form. Patients are followed until the time of death.

NOTE: *If a patient is not available for the scheduled home visit, the interview will take place over the phone; if a patient is hospitalized or transferred to the inpatient hospice facility, the patient interview will take place there.

* Primary caregiver assessment**: At baseline, primary caregivers complete a demographic survey, a Pain Assessment Form, the Pain Communication Survey, Caregiver Self-Efficacy in Pain Management Scale (CSEPMS), the Caregiver Pain Management Questionnaire (CPMQ), and the Stressful Caregiver Adult Reactions to Experiences of Dying (SCARED). Caregivers are then interviewed by the study nurse using the Pain Assessment Form as a guideline. Follow-up data from caregivers is obtained through a daily diary, interviews, and structured surveys. Primary caregivers complete the Pain Assessment Form daily and are instructed to provide their assessment of the patient's pain. In addition, caregivers are interviewed daily by a study nurse, who reviews the daily Pain Assessment Form and obtains detailed information regarding the adequacy of patient pain control, side effects of medication, barriers to pain control, and caregiver concerns and burdens. Primary caregivers also complete CSEPMS, CPMQ, and SCARED questionnaires at the end of weeks 1, 2, and 4 as part of follow-up. Primary caregivers are contacted after the patient's death to assess pain control at the time of death.
* Secondary caregiver assessment: At baseline, secondary caregivers complete the same baseline evaluation as primary caregivers over the phone. They complete the Pain Assessment Form weekly and the CSEPMS, CPMQ, and SCARED questionnaires at the end of weeks 1, 2, and 4. Secondary caregivers also undergo a post-mortem interview based on the Pain Assessment Form.
* Chart review: Chart review is conducted by the research Nurse after a patient's death. Cancer and cancer-related treatment are obtained and documentation about pain management is recorded. From the time of study entry, all staff notes are reviewed to document: pain assessment, calls to physicians or other support personnel (including pharmacy calls), identified barriers to pain control, and treatment modifications (including medications to treat side effects).

NOTE: **Patients and primary caregivers are interviewed independently.

ELIGIBILITY:
Inclusion Criteria:

Patient eligibility includes:

* Alive Hospice outpatient
* Diagnosis of carcinoma
* Pain requiring fixed dose opioids
* Age > 21 years
* Not pregnant or lactating
* Willing and able to sign informed consent -Able to speak/comprehend English

Caregiver eligibility will include:

* Caregiver for an Alive Hospice patient
* Willing and able to sign informed consent
* Able to speak/comprehend English

Exclusion Criteria:

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in Alive hospice who have pain and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Description of standard pain management methods and outcomes in the hospice setting | date on study to death

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States